CLINICAL TRIAL: NCT00386256
Title: Home Based Telerehabilitation for Deconditioned Older Adults
Brief Title: Home Telerehabilitation for Deconditioned Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Model: Parallel | Masking: None
Other Study IDs: E4204-R; NCT00929149 (obsolete NCT alias)
Record Dates: First submitted 2006-10-06; First posted 2006-10-11 (Estimated); Results first posted 2014-08-15 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-08

CONDITIONS: Osteoarthritis
Keywords: telehealth; telerehabilitation; deconditioning; exercise
MeSH Terms: conditions — Osteoarthritis; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Health Buddy outpatient (Experimental): Received home telehealth monitoring by Health Buddy
  Interventions: Device: Health Buddy, Home telehealth technology
- Telephone outpatient (Experimental)
  Interventions: Other: Telephone counseling
- health buddy inpatient (Experimental)
  Interventions: Device: Health Buddy, Home telehealth technology
- telephone inpatient (Experimental)
  Interventions: Other: Telephone counseling

INTERVENTIONS:
Device: Health Buddy, Home telehealth technology — Exercise questions, educational messages, and clinical reminders have been programmed into the home telehealth technology and are administered daily via the Health Buddy(R) to evaluate the program's feasibility based on adherence rates, program completion rates, and safety.
  Arms: Health Buddy outpatient; health buddy inpatient
Other: Telephone counseling
  Arms: Telephone outpatient; telephone inpatient

SUMMARY:
The purpose of this study is to develop a home exercise program for patients 60 years of age and over who are deconditioned following their discharge from the hospital, or recruited from GLA outpatient clinics. The program will be designed to monitor and improve patients' exercise behavior through the use of home technology, such as text messaging monitors.

DETAILED DESCRIPTION:
The aim of this study is to develop and determine the feasibility of implementing a home exercise and functional status monitoring telerehabilitation program, known as TEL-REHAB, for older adults 60 years of age and over who are deconditioned following their discharge from the inpatient setting, or recruited from GLA outpatient clinics. Deconditioning is a modifiable risk factor for preventing institutionalization of frail elderly patients who would otherwise be able to live independently. Home exercise programs are an effective intervention to reduce the risk, but patient compliance with home exercise programs, and assessments of patients during home exercise programs, are barriers to achieving maximal benefits. Face-to-face visits with physical medicine professionals are an effective means to perform these functions, but are problematic because of professional time impacts and patient transportation problems. A TEL-REHAB program will empower these patients to take responsibility for their own health by providing ongoing communication with a healthcare provider. In this way, telerehabilitation may assist older adults to remain independent in their homes as long as possible.

ELIGIBILITY:
Inclusion Criteria:

* acute decline in functional status while hospitalized as reported by the patient
* physically inactive outpatients (exercise less than 30 min/day, 3 d/wk)
* ability to hear and communicate via telephone
* ability to read a video or text monitor
* ability to manually operate the technology
* have a working telephone and power source
* willingness to use the TEL-REHAB technology

Exclusion Criteria:

* does not speak English
* poor cognition as determined by the Mini-Cog
* non-ambulatory
* had a stroke, myocardial infarction, hip fracture, or total hip or knee replacement within the prior 6 months

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2006-10; Primary Completion 2008-05 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy D. Harada, PhD MPA, Principal Investigator — VA Greater Los Angeles Healthcare System, West LA
Locations (1):
- VA Greater Los Angeles Healthcare System, West LA, West Los Angeles, California, United States

REFERENCES:
- [Derived] Harada ND, Dhanani S, Elrod M, Hahn T, Kleinman L, Fang M. Feasibility study of home telerehabilitation for physically inactive veterans. J Rehabil Res Dev. 2010;47(5):465-75. doi: 10.1682/jrrd.2009.09.0149. PMID 20803390

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from both the inpatient and outpatient settings of a large urban academic VA hospital. Potential participants were recruited through referrals from physicians, case managers, and social workers, participant recruitment fairs, and flyers posted around the hospital.
Groups:
- Health Buddy Outpatient: Health Buddy(R), Home telehealth technology : Exercise questions, educational messages, and clinical reminders have been programmed into the home telehealth technology and are administered daily via the Health Buddy(R) to evaluate the program's feasibility based on adherence rates, program completion rates, and safety.
Period: Overall Study
Arm/Group | Health Buddy Outpatient | Telephone Outpatient | Health Buddy Inpatient | Telephone Inpatient
Started | 16 | 15 | 4 | 3
Completed | 16 | 15 | 4 | 3
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Health Buddy Outpatient: Received Health Buddy, recruited from outpatient setting
- Telephone Outpatient: Received telephone counseling, recruited from outpatient setting
- Health Buddy Inpatient: Received Health Buddy, recruited from inpatient setting
- Telephone Inpatient: Received telephone counseling, recruited from inpatient setting
- Total: Total of all reporting groups
Arm/Group | Health Buddy Outpatient | Telephone Outpatient | Health Buddy Inpatient | Telephone Inpatient | Total
Number analyzed (Participants) | 16 | 15 | 4 | 3 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 0 | 0 | 2
  >=65 years | 15 | 14 | 4 | 3 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.9 (7.9) | 65 (6.1) | 78 (4.7) | 76 (7.5) | 72.2 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 16 | 15 | 4 | 3 | 38
Region of Enrollment [Number; unit: participants]
  United States | 16 | 15 | 4 | 3 | 38

OUTCOME MEASURES:

1. Primary Outcome: Exercise Adherence
Description: An 11-week exercise adherence rate was calculated by dividing the total number of days that the participant reported exercising by 77 days and multiplying by 100. This first calculation estimated the exercise adherence rate for the full intervention period regardless of participant dropout. Eleven weeks rather than 12 weeks was used in the denominator because subjects received their HB units some time during the first week of study enrollment and may have missed some days during this first week.
Time Frame: at monthly intervals, for 3-months
Measure: Mean (Standard Deviation); unit: percentage of days adhered
Arm/Group | Health Buddy Outpatient | Telephone Outpatient | Health Buddy Inpatient | Telephone Inpatient
Number analyzed (Participants) | 16 | 15 | 4 | 3
percentage of days adhered | 57.4 (24.9) | 32.1 (22.7) | 56.2 (15.6) | 35.1 (20.0)
Statistical Analysis 1: Comparison: Health Buddy Outpatient vs Telephone Outpatient vs Health Buddy Inpatient vs Telephone Inpatient; Statistical analyses included descriptive statistics to assess demographic and medical characteristics, safety, text messaging or phone adherence, exercise adherence, and patient satisfaction. T-tests were used to determine significant differences between the HB text messaging and telephone groups (with inpatients and outpatients combined within each group). All analyses were conducted using SPSS version 14.0 for Windows; Test type: Superiority or Other; p < .05, t-test, 2 sided

2. Primary Outcome: HB/Phone Adherence
Description: An 11-week text messaging or phone adherence rate was calculated by dividing the number of response days via the HB or phone divided by 77 days and multiplied by 100. This first calculation estimated the text messaging or phone adherence rate for the full intervention period regardless of participant dropout. Eleven weeks rather than 12 weeks was used in the denominator because subjects received their HB units some time during the first week of study enrollment and may have missed some days during this first week.
Time Frame: Monthly over 3 months
Measure: Mean (Standard Deviation); unit: percentage of days adhered
Arm/Group | Health Buddy Outpatient | Telephone Outpatient | Health Buddy Inpatient | Telephone Inpatient
Number analyzed (Participants) | 16 | 15 | 4 | 3
percentage of days adhered | 64.7 (29.7) | 36.3 (24.2) | 70.1 (26.3) | 43.7 (25.8)
Statistical Analysis 1: Comparison: Health Buddy Outpatient vs Telephone Outpatient vs Health Buddy Inpatient vs Telephone Inpatient; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < .05, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Health Buddy Outpatient | Telephone Outpatient | Health Buddy Inpatient | Telephone Inpatient
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/15 | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 4/16 | 1/15 | 3/4 | 0/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Health Buddy Outpatient (N=16) | Telephone Outpatient (N=15) | Health Buddy Inpatient (N=4) | Telephone Inpatient (N=3)
Chest tightness (General disorders) | 2 (4) | 1 (1) | 2 (2) | 0 (0)
Dizziness (General disorders) | 2 (4) | 0 (0) | 2 (2) | 0 (0)
Trips/Falls (General disorders) | 4 (4) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Intervention was developed on a male Veteran population, direct comparisons between groups were formed based on the participant's preference, exercise adherence was based on participants' self reports, small convenience sample.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes